CLINICAL TRIAL: NCT03799900
Title: A Two-part, Single-dose, Randomized, Double-blind, Placebo and Active-Controlled Crossover Study to Evaluate the Abuse Potential of Rapastinel in Healthy, Non-dependent, Adult Recreational Polydrug Users
Brief Title: Assessment of Abuse Potential of Rapastinel in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RAP-PK-12
Record Dates: First submitted 2018-11-15; First posted 2019-01-10 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Human Abuse Potential
MeSH Terms: interventions — GLYX-13 peptide; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1, Cohort 1: Ketamine Low Dose (Experimental): Some participants will be administered a single IV dose of ketamine on Day 1.
  Interventions: Drug: Ketamine
- Part 1, Cohort 1: Placebo (Placebo Comparator): Some participants will be administered a single IV dose of placebo on Day 1.
  Interventions: Drug: Placebo
- Part 1, Cohort 2: Ketamine Medium Dose (Experimental): Some participants will be administered a single IV dose of ketamine on Day 1.
  Interventions: Drug: Ketamine
- Part 1, Cohort 2: Placebo (Placebo Comparator): Some participants will be administered a single IV dose of placebo on Day 1.
  Interventions: Drug: Placebo
- Part 1, Cohort 3 (Optional): Ketamine High Dose (Experimental): Optional: some participants will be administered a single IV dose of ketamine on Day 1.
  Interventions: Drug: Ketamine
- Part 1, Cohort 3 (Optional): Placebo (Placebo Comparator): Optional: some participants will be administered a single IV dose of placebo on Day 1.
  Interventions: Drug: Placebo
- Part 2, Qualification Phase: Ketamine (Experimental): Participants will receive IV ketamine on Day 1 and placebo on Day 2 in a randomized crossover manner.
  Interventions: Drug: Ketamine
- Part 2, Qualification Phase: Placebo (Placebo Comparator): Participants will receive IV ketamine on Day 2 and placebo on Day 1 in a randomized crossover manner.
  Interventions: Drug: Placebo
- Part 2, Treatment Phase: Rapastinel Low Dose (Experimental): Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel
- Part 2, Treatment Phase: Rapastinel Medium Dose (Experimental): Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel
- Part 2, Treatment Phase: Rapastinel High Dose (Experimental): Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel
- Part 2, Treatment Phase: Ketamine (Active Comparator): Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Interventions: Drug: Ketamine
- Part 2, Treatment Phase: Placebo (Placebo Comparator): Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — During the Treatment Phase in Part 2, participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Arms: Part 2, Treatment Phase: Rapastinel High Dose; Part 2, Treatment Phase: Rapastinel Low Dose; Part 2, Treatment Phase: Rapastinel Medium Dose
Drug: Ketamine — Part 1
  Part 2, Qualification Phase:
  Participants will be administered single IV doses of ketamine and placebo in a randomized crossover manner
  Part 2, Treatment Phase:
  Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Arms: Part 1, Cohort 1: Ketamine Low Dose; Part 1, Cohort 2: Ketamine Medium Dose; Part 1, Cohort 3 (Optional): Ketamine High Dose; Part 2, Qualification Phase: Ketamine; Part 2, Treatment Phase: Ketamine
Drug: Placebo — Part 1
  Part 2, Qualification Phase:
  Participants will be administered single IV doses of ketamine and placebo in a randomized crossover manner
  Part 2, Treatment Phase:
  Participants will be administered single IV doses of rapastinel, ketamine, and placebo in a randomized crossover manner.
  Arms: Part 1, Cohort 1: Placebo; Part 1, Cohort 2: Placebo; Part 1, Cohort 3 (Optional): Placebo; Part 2, Qualification Phase: Placebo; Part 2, Treatment Phase: Placebo

SUMMARY:
Based on the pharmacological class of rapastinel, this study will be conducted to evaluate the abuse potential of single doses of rapastinel as compared with ketamine, a NMDAR antagonist that is a Schedule III dissociative anesthetic, and placebo in recreational polydrug users.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a current recreational polydrug user
* Have a supine systolic blood pressure (BP) ≥ 95 mm Hg and ≤ 145 mg Hg, or supine diastolic BP ≥ 50 mm Hg and ≤ 90 mm Hg at the Screening Visit.
* Have negative test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, alcohol, oxycodone and other opioids, and phencyclidine at any admission
* Able, as assessed by the investigator, and willing to follow study instructions and likely to complete all required study visits

Exclusion Criteria:

* Evidence of drug or alcohol dependence (excluding nicotine and caffeine) within the past 2 years
* Suicidal risk based on the opinion of the principal investigator (or appropriately trained designee)
* History of violent or psychotic behavior when taking psychedelic drugs, or unwilling to take a drug that might alter perception in a controlled setting
* Have taken or require concomitant treatment with any CNS depressants, or cannot safely discontinue these medications within 14 days (or 5 half-lives, whichever is longer) before study treatment administration
* Previously participated in an investigational study of rapastinel.
* Participation in any other clinical investigation using an experimental drug within 30 days, 5 half-lives or twice the duration of the biological effect of the study treatment (whichever is longer), prior to study treatment administration or is concurrently enrolled in any clinical trial, judged not to be scientifically or medically compatible with this study
* Consumption of alcohol within 72 hours before administration of study treatment
* Breastfeeding
* Unable to refrain from consuming caffeine or xanthine-containing compounds such as tea, coffee, soft drinks, energy sports drinks or chocolate (more than 48 oz/day) from 48 hours before administration of study treatment.
* Have consumed dietary supplements or other foods or beverages that may affect various drug metabolizing enzymes and transporters (eg, grapefruit, grapefruit juice, grapefruit-containing beverages), vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats within 14 days prior to dosing or unable to refrain from consumption during the study.
* The ability to tolerate IV ketamine as judged by the Investigator, based on available safety data, as well as pharmacodynamic data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Maximum effect (Emax) for "At this Moment" Drug Liking visual analog scale (VAS). | Treatment Phase: Pre-dose and up to 24 hours post-dose
  The drug liking VAS measures the participant's liking for the drug and is scored from 0 to 100, with 0 reflecting "Strong disliking" and 100 reflecting "Strong liking".

SECONDARY OUTCOMES:
Maximum effect (Emax) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Minimum effect (Emin) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Time to Emax (TEmax) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Time to Emin (TEmin) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Time averaged area under the effect curve (TA_AUE) | Treatment Phase: Hour 0 and up to 24 Hours post-dose
Maximum plasma drug concentration (Cmax) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration (AUClast) | Treatment Phase: Pre-dose and up to 24 hours post-dose
Adverse events | Part 1: 6 weeks, Part 2: 9 weeks
Proportion of abnormal electrocardiograms | Part 1: 6 weeks, Part 2: 9 weeks
Columbia-Suicide Severity Rating Scale | Part 1: 6 weeks, Part 2: 9 weeks
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (least severe) to 5 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Fang Su, Study Director — Allergan
Locations (1):
- Vince and Associates Clinical Research Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided